CLINICAL TRIAL: NCT03057717
Title: The Effect of Antenatal Corticosteroids on the Fetal Thymus - a Possible Role in Fetal Immune
Brief Title: The Effect of Antenatal Corticosteroids on the Fetal Thymus - a Possible Role in Fetal Immune Programming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-189
Record Dates: First submitted 2017-02-03; First posted 2017-02-20 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Preterm Labor; Fetal Glucocorticoid Exposure
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Other): All participants in the study will have fetal thymus size measured using ultrasound.
  Interventions: Other: 2D ultrasound assessment

INTERVENTIONS:
Other: 2D ultrasound assessment — 2D ultrasound assessment of fetal thymus size with measurements of the maximum transverse diameter and thymus perimeter

SUMMARY:
Administration of corticosteroids is standard practice for pregnant patients at risk of preterm labour to reduce the risk of neonatal respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis and neonatal mortality. However, there is an unknown effect of antenatal steroids on both fetal and neonatal immune function. The purpose of this study is to demonstrate the effect of antenatal steroids on the size of the fetal thymus gland.

DETAILED DESCRIPTION:
Women with a singleton pregnancy in the twenty-forth to thirty-fourth week of gestation who are at risk for preterm labour, requiring the administration of Betamethasone twelve milligrams intramuscularly every twenty-four hours for two doses will be included in this study along with an equal number of gestational-age matched controls not at risk for preterm delivery and therefore not requiring the administration of Betamethasone. A 2-D ultrasound assessment of the fetal thymus size with measurements of the maximum transverse diameter and thymus perimeter in the three-vessel view will be performed as a baseline measurement within 36 hours of the administration of the first dose of corticosteroids. For each patient enrolled, a gestational-age matched control will have a similar ultrasound assessment. These measurements will be repeated 2 weeks after the first baseline ultrasound, and then only patients who received corticosteroids will have subsequent ultrasound measurements every 2 weeks until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy in the twenty-forth to thirty-fourth week of gestation who are at risk for preterm labour, requiring the administration of Betamethasone twelve milligrams intramuscularly every twenty-four hours for two doses will be included in this study along with an equal number of gestational-age matched controls not at risk for preterm delivery and therefore not requiring the administration of Betamethasone.

Exclusion Criteria:

* chronic use of steroids during pregnancy for other indications
* delivery less than 1 week from enrollment
* confirmed chorioamnionitis or preterm premature rupture of membranes.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 86 (Actual)
Dates: Start 2010-08-20 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Fetal Thymus Size | 24 weeks gestation to delivery
  Fetal thymus size for pregnant women given Betamethasone compared to fetal thymus size for pregnant women not given Betamethasone

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No